CLINICAL TRIAL: NCT05499234
Title: Effects of Different Local Anesthetic Concentrations With Epidural Tap Method for Labor Analgesia
Brief Title: Epidural Tap in Labor Analgesia FOR LABOR ANALGESIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Pelin Karaaslan, Professor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KARAASLANP
Record Dates: First submitted 2022-08-02; First posted 2022-08-12 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Labor Pain
Keywords: labor analgesia; dural tap; concentration
MeSH Terms: conditions — Labor Pain | interventions — Meperidine; Acetaminophen

STUDY DESIGN:
Intervention Model Description: 70 ASA II primigravid women with cervical dilatation between 4-6 cm and demanding epidural analgesia during spontaneous vaginal delivery
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and the medical staff administrating epidural drugs will not be told about the concentration. Because volumes will be same, they would not predict which group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High concentration (Experimental): Epidural analgesia with 20 mL of 0.125% bupivacaine + 2 mcg/mL fentanyl solution
  Interventions: Drug: Dolantin; Drug: Paracetamol
- Low concentration (Experimental): Epidural analgesia with 20 mL of 0.0625% bupivacaine + 2 mcg/mL fentanyl solution
  Interventions: Drug: Dolantin; Drug: Paracetamol

INTERVENTIONS:
Drug: Dolantin — If VAS score is more than 4 even after additional dose, use dolantin 1 mg/kg
  Other Names: Meperidin
Drug: Paracetamol — If VAS score is more than 4 even after dolantin 1 mg/kg, 10 mg/kg paracetamol IV
  Other Names: Parol

SUMMARY:
The dural epidural tap method is performed by creating a dural perforation with a spinal needle placed through epidural needle, followed by placement of a catheter into the epidural space. No medications are administered through spinal needle. This prospective, randomized study includes 70 ASA II primigravid women with cervical dilatation between 4-6 cm and demanding epidural analgesia during spontaneous vaginal delivery.In the first group, 20 mL of 0.125% bupivacaine + 2 mcg/mL fentanyl solution and in the second group, 20 mL of 0.0625% bupivacaine + 2 mcg/mL fentanyl solution was administered as the first dose through the epidural catheter. Then, the visual analog scale (VAS) score was aimed to be below 4 in both groups.

DETAILED DESCRIPTION:
This prospective, randomized study includes 70 ASA II primigravid women with cervical dilatation between 4-6 cm and demanding epidural analgesia during spontaneous vaginal delivery. Participants with pregnancy-related diseases (such as gestational hypertension, gestational diabetes, preeclampsia) and contraindications for neuraxial block (infection, coagulation disorder, severe hypovolemia, sepsis, neurological deficit, cardiac valve stenosis or hypertrophic obstructive cardiomyopathy) will be excluded from the study. Women with fetal malpresentation and fetal anomaly will also be excluded.

Participants will randomly be divided into 2 equal groups. Immediately before epidural placement, subjects will be marked a VAS score during an active contraction. All subjects will have an intravenous catheter placed and be monitored with NST, noninvasive blood pressure and pulse oximetry.

The epidural space will be identified by a loss of resistance technique to saline. CSF flow will be observed at L3-L4 or L4-L5 level by puncturing the dura with a 27 G needle before inserting the epidural catheter. A combined spinal epidural set with 18 G Tuohy needle will be used in both groups. In the first group, 20 mL of 0.125% bupivacaine + 2 mcg/mL fentanyl solution and in the second group, 20 mL of 0.0625% bupivacaine + 2 mcg/mL fentanyl solution will be administered as the first dose through the epidural catheter. Then, the visual analog scale (VAS) score will be aimed to be below 4 in both groups. Patients with a VAS score of 4 or higher 15 minutes after the first dose received, an additional 10 mL dose of the same solution will be given. An additional 10 mL dose also will be administered when the VAS score is 4 or higher until crowning.

Before the epidural catheter placed; age, weight, height, blood pressure of the participants, gestational week, use of oxytocin during delivery, cervical dilatation amount before the procedure and fetal heart rate will be recorded. After each dose of administration, whether maternal hypotension, fetal bradycardia, pruritus, nausea-vomiting or motor block development will be monitored. The total amount of drug administered through the epidural catheter, the time between applications, and the number of bolus doses administered will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA II primigravid women
* with cervical dilatation between 4-6 cm, demanding epidural analgesia during spontaneous vaginal delivery

Exclusion Criteria:

* Participants with pregnancy-related diseases

  * gestational hypertension
  * gestational diabetes
  * preeclampsia/ celmpsia
* contraindications for neuraxial block

  * infection
  * coagulation disorders
  * severe hypovolemia
  * sepsis
  * neurological deficit
  * cardiac valve stenosis or hypertrophic obstructive cardiomyopathy
* Women with fetal malpresentation and fetal anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Change the need of bupivacaine for epidural analgesia. | In an hour
  primary aim of this study is to achieve Numeric Pain Rating Scale scores equal to or below 4 via different bupivacaine concentrations. More than 4 is bad and unacceptable

SECONDARY OUTCOMES:
Complication comparison | 2 days
  measure the number of treatment related complications and compare these measurements between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Uçar, Principal Investigator — Medipol University; Emine Uzunoğlu, Study Chair — Medipol University; Pelin Karaaslan, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Bağcılar, Turkey (Türkiye)

REFERENCES:
- [Derived] Ucar FP, Danisan HG, Omur B, Alici HA, Karaaslan P. Effects of different bupivacaine concentrations with dural puncture epidural technique for labor analgesia: a prospective randomized controlled trial. BMC Anesthesiol. 2025 Nov 26;25(1):590. doi: 10.1186/s12871-025-03486-0. PMID 41299385